CLINICAL TRIAL: NCT05390268
Title: Mobile App-assisted Behavioral Treatment (MA-BT) in Children and Adolescents With a Chronic Tic Disorder. Randomized Clinical Trial Evaluating Treatment Response and Satisfaction
Brief Title: Mobile App-assisted Behavioral Treatment in Children and Adolescents With Tics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Judith Becker Nissen, associate professor, phd, senior doctor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-16-02-355-21
Record Dates: First submitted 2022-05-01; First posted 2022-05-25 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Tic Disorders
Keywords: tics; children; adolescents; Mobile app-assisted behavioral treatment
MeSH Terms: conditions — Tic Disorders; Tics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor is not involved in the treatment of the patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digital tic training (Experimental): The active treatment including apps released for every session
  Interventions: Behavioral: Mobile app-assisted behavioral treatment
- digital tic learner (Active Comparator): The control arm including apps released in the first session
  Interventions: Other: Mobile app-assisted psychoeducation

INTERVENTIONS:
Behavioral: Mobile app-assisted behavioral treatment — The app-assisted training group has access to a newly developed app in which they are taught how to handle tics. A new app session is released at each new treatment session and the content of the app videos is comparable to the information and training at face-to-face individual treatment, as defined by the manual "Niks to Tics"[
  Arms: digital tic training
Other: Mobile app-assisted psychoeducation — The app-assisted educational group has access to a newly developed app in which they receive psychoeducation on tics.
  Arms: digital tic learner

SUMMARY:
Chronic tic disorders are neurodevelopmental disorders affecting 0.5-1% of children and adolescents. Tics present as sudden, rapid, repetitive non-rhythmic movements or vocalizations or a combination. Tics may be extremely distressing in a child's life, but the severity of tics is often variable. The group of children/ adolescents with tic disorders are heterogenous when it comes to symptom presentation, comorbid conditions and social status. This places great demands on professionals to offer the right treatment at the right time. The aim of the current project is to make optimal tics training more accessible, including for patients managed in primary care, to make optimal treatment available in the immediate environment, and to ensure increased adherence to treatment.

As part of this project, an app has been developed and the study aims to evaluate mobile app-assisted behavioral treatment as an efficient and feasible approach that may be a valuable tool together with other treatment approaches. The mobile app-assisted training is based on the manual "Niks til Tics", which describes training with a combination of Habit Reversal Training (HRT) and Exposure Response Prevention (ERP) over eight sessions, and a booster session. Both HRT and ERP are known to be effective treatments of tics.

In this project a randomized controlled superiority trial evaluates the effect of app-assisted training versus an educational approach. Participants are randomized to manualised treatment combining HRT and ERP as app-assisted training, or to psychoeducation. The participants are included according to the same criteria as in a pilot trial, and primary outcome measure is YGTSS at session 8. Furthermore, the change in tics intensity from the first contact to baseline will be included as to evaluate the effect of being admitted and examined at the hospital.

This project contributes to increased knowledge about tics and tic treatment especially treatment using digital based interventions. An app has been developed for this project and the hypothesis is that a mobile app-assisted tic training program requiring minimal hospital contacts is superior to app-based psychoeducation alone, which is the most likely intervention that these patients will be offered.

This registration encompasses a project that collects information/data for multiple publications. As such, a number of publications are planned including a description of acute outcome, potential predictors, and longterm treatment effect

ELIGIBILITY:
Inclusion Criteria:

* a primary diagnosis of a chronic motor/vocal tics disorder including Tourette syndrome according to the WHO ICD-10 diagnostic criteria and Statistical Manual of Mental Disorders
* a total tic score higher than 13 on the Yale Global Tic Severity Scale (YGTSS), or above a tic score of 9, if only motor or vocal tics are present

Exclusion Criteria:

* psychotic disorder
* primary severe depression
* suicidal ideation or attempts
* primary severe eating disorder
* IQ below 70 (mental retardation)
* participation in tic training based on HRT/ERP treatment within 6 months

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of baseline Yale Global Tic Severity Scale (YGTSS) at 5 weeks, 15 weeks, 23 weeks, 75-96 weeks | Baseline, 5 weeks, 15 weeks, 23 weeks, 75-96 weeks
  YGTSS - a clinician-administered semi-structured interview including a checklist of all tic symptoms

SECONDARY OUTCOMES:
Change of baseline premonitory urge scale (PUTS) | Baseline, 5 weeks, 15 weeks, 23 weeks, 75-96 weeks
  PUTS is a short self-reporting scale with nine items
Change of baseline beliefs about tics scale (BATS) | Baseline, 5 weeks, 15 weeks, 23 weeks, 75-96 weeks
  BATS is a self-reporting scale with 20 items
Change of baseline parent and child self-evaluating questionnaire | Baseline, 5 weeks, 15 weeks, 23 weeks, 75-96 weeks
  Based on PTQ - a parent evaluating questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Per Thomsen, Phd, Study Chair — Department of Child and Adolescent Psychiatry, Aarhus University Hospital, Psychiatry, Aarhus, Denmark
Locations (1):
- AarhusUH, Aarhus N, Risskov, Denmark

IPD SHARING:
Plan to Share IPD: No